CLINICAL TRIAL: NCT07022548
Title: Prospective Study Evaluating the Prevalence of Intestinal Dysfunction in Hematology Patients Hospitalized in Intensive Care for Sepsis or Septic Shock
Brief Title: Prospective Study Evaluating the Prevalence of Intestinal Dysfunction
Acronym: DIR-H
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/060/OB; N° IDRCB : 2023-A00552-43 (Other: ANSM)
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-01

CONDITIONS: Intestinal Inflammation
Keywords: sepsis/septic shock; prevalence
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — fecal and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient admitted to intensive care for sepsis or septic shock with malignant hematological disease
- Patient admitted to intensive care for sepsis or septic shock without malignant hematological diseas

SUMMARY:
The intestinal tract has multiple functions within the body beyond its primary function of nutrient absorption. It acts as a true barrier protecting the body from living microorganisms and antigens in the intestinal lumen. Impairment of any component of the intestinal barrier results in nutrient malabsorption, an altered local digestive immune response, and increased intestinal permeability.

The primary function of this barrier is to limit the access of the contents of the intestinal lumen, which particularly includes the bacterial components of the microbiota, to the internal environment and the circulation. This physical barrier function is provided by a monolayer of epithelial cells, closely connected to each other by intercellular junctions (tight junctions, adherens and desmosomes, as well as by the mucus which covers the apical surface of the cells, the constituents of which, mucins, are secreted by the goblet cells. The term intestinal barrier is also used in a broader sense including a protective role against the invasion of environmental pathogens, while allowing toleranSepsis-associated intestinal failure is often underestimated, yet it is found in 20 to 60% of ICU (Intensive Care Unit)vpatients. However, its prognosis is poorly documented. For example, there is no consensus definition of this dysfunction or validated biomarkers for rapid assessment. Consequently, it does not appear in most prognostic scores (SOFA, IGS2, etc.).

Intestinal permeability, a risk factor for bacterial translocation when elevated, is increased in ICU (Intensive Care Unit) patients and associated with multiorgan failure system (MODS), particularly in cases of intestinal fasting. However, there is currently no validated marker of acute intestinal failure in intensive care or intensive care.ce towards commensal flora and foods.

DETAILED DESCRIPTION:
Several markers of intestinal response have been studied and are still in the research field due to a lack of conclusive work on their impact.

Clinically, both in post-weaning children and in adults, citrullinemia (citrulline deficiency) is well established as a sensitive and specific indicator of functional absorptive enterocyte mass.

Fecal calprotectin is already used as a marker of neutrophil-mediated inflammation in inflammatory bowel disease.

A recent controlled observational study of 165 patients investigated serum calprotectin as a prognostic marker in sepsis patients hospitalized in critical care. The authors found a significant increase in serum calprotectin concentration in sepsis patients compared to control patients. Furthermore, it would appear that a high level of calprotectin upon admission to intensive care is a significant risk factor for long-term mortality.

Finally, in patients with sepsis, serum zonulin levels are elevated, which promotes bacterial translocation via the epithelium and thus bacteremia.

The risk of infection in immunocompromised patients is a therapeutic challenge due to its adverse prognostic impact. Sepsis-related mortality is higher (relative risk = 1.62) in immunocompromised patients. One of the mechanisms of sepsis in these patients is gastrointestinal bacterial translocation due to the gastrointestinal cytotoxicity of chemotherapy, microbiota alterations via antibiotic therapy, and low perfusion rates.

This study aims to assess the prevalence of intestinal inflammation in a population of patients with malignant hematological diseases undergoing treatment and admitted to intensive care for sepsis-septic shock. These patients are exposed to cytotoxic chemotherapies that attack the intestinal mucosa, making it more permeable and thus being the source of digestive translocations of bacteria from the intestinal microbiota into the bloodstream. In the absence of validated threshold values in the literature to define intestinal inflammation based on fecal calprotectin levels, it is necessary to have a control population also affected by sepsis but not carrying malignant hematological disease.

ELIGIBILITY:
Inclusion Criteria:

Population with hematologic malignancy

* Patients over 18 years of age
* Suffering from hematologic malignancy
* Admitted to intensive care for sepsis or septic shock according to sepsis definition 3:

  * Sepsis: organ dysfunction (SOFA > or = 2) related to a host response to infection
  * Septic shock: sepsis with acute circulatory failure and metabolic abnormalities (serum lactate > 2 mmol/L) and vasopressors
* Patients who have read and understood the information letter and do not object to participating in the study
* Affiliated with or beneficiary of a social security scheme.

Control population

- Patient aged over 18

Admitted to intensive care for sepsis or septic shock according to the sepsis definition 3:

* Sepsis: organ dysfunction (SOFA > or = 2) related to a host response to infection
* Septic shock: sepsis with acute circulatory failure and metabolic abnormalities (serum lactate > 2 mmol/L) and vasopressors

  * Patient who has read and understood the information letter and does not object to participating in the study
  * Member of or beneficiary of a social security scheme

Exclusion Criteria:

For the control group and those with hematologic malignancies:

* Patient refusal
* Pregnant, parturient, or breastfeeding woman
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection/guardianship or curatorship
* Person who does not understand or speak French
* Moribund
* Limitations of active therapies (LATA) established upon admission
* Hospitalization in intensive care > 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients with malignant haemopathy admitted for sepsis or septic shock in intensive care and a control population of 40 patients admitted to intensive care for sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of intestinal inflammation | 72 hours after enrollment visit
  To assess the prevalence of intestinal inflammation defined by the fecal calprotectin level on admission (<72 hours) in patients with malignant hematological disease admitted to intensive care for sepsis or septic shock.

SECONDARY OUTCOMES:
Prevalence of intestinal hyperpermeability | 72 hours after enrollment visit
  To assess the prevalence of intestinal hyperpermeability defined by the plasma level of zonulin taken between admission and H72 in patients with malignant haemopathy admitted to intensive care for sepsis or septic shock (compared to the control population also suffering from sepsis but not carrying malignant haemopathy)
Prevalence of intestinal hyperpermeability | 72 hours after enrollment visit
  To assess the prevalence of intestinal hyperpermeability defined by the fecal zonulin level on admission taken between admission and H72 in patients with malignant haemopathy admitted to intensive care for sepsis or septic shock (compared to the control population)
Integrity of intestinal tissue | 72 hours after enrollment visit
  To assess the integrity of intestinal tissue defined by the level of plasma IFABP collected between admission and H72 in patients with malignant haemopathy admitted to intensive care for sepsis or septic shock (compared to the control population)
Impact of intestinal dysfunction on the occurrence of digestive intolerance | month 6
  Assess the impact of intestinal dysfunction on the occurrence of digestive intolerance: vomiting, diarrhea, constipation, occlusive syndrome
Impact of intestinal dysfunction on mortality | month 6
  Evaluation of the impact of intestinal dysfunction on mortality in intensive care and hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne FT TAMION, Professor, Principal Investigator — University Hospital, Rouen
Locations (1):
- Médecine Intensive Réanimation, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.